CLINICAL TRIAL: NCT01857648
Title: Physical Activity Promotion in the Brazilian Primary Health Care Using Community Health Workers Counseling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Alex Antonio Florindo, Ph.D., University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2009/14119-5
Record Dates: First submitted 2013-05-15; First posted 2013-05-20 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-05

CONDITIONS: Physical Activity
Keywords: Physical Activity; Health Promotion; Primary Health Care; Intervention Studies; Public health Practice
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical activity counseling (Experimental): Home visits including physical activity promotion by the trained Community Health Workers.
  Interventions: Other: Physical activity counseling
- Control (No Intervention): Control group.

INTERVENTIONS:
Other: Physical activity counseling — Home visits including physical activity promotion by the trained Community Health Workers.
  Arms: Physical activity counseling

SUMMARY:
The aim of this study is to test a methodology of counseling on physical activity among Community Health Workers working within primary health care in Brazil.

DETAILED DESCRIPTION:
This is an intervention study conducted with 176 people attended by two Primary Health Units in the city of São Paulo, Brazil. The intervention group received home visits of Community Health Workers trained on counseling on physical activity promotion. These workers received a course of 12 hours aimed to improve their knowledge and attitude about physical activity promotion. Evaluations will be done at the study baseline and 6 months after the beginning. The primary outcome is the population leisure-time and transport-related physical activity level.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or more
* To be registered in the Brazilian public health system

Exclusion Criteria:

* Health problem or disease that would make the individual incapable of practice physical activity
* Cognitive problem or disease that would not allow the individual from answering the questionnaire alone
* To have plans to move house over the six-months subsequent period
* Being pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2011-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline leisure-time and transport-related physical activity at 6 months | 6 months
  Measured in minutes per week

SECONDARY OUTCOMES:
Change from baseline self-rated health at 6 months | 6 months
Change from baseline stage of behavior change at 6 months | 6 months
Change from baseline barriers to physical activity practice at 6 months | 6 months
Change from baseline Community Health Workers's counseling on physical activity at 6 months | 6 months
Change from baseline Community Health Workers's knowledge about physical activity promotion at 1 month | 1 month
Change from baseline Community Health Workers's knowledge about physical activity promotion at 5 months | 5 months
Change from baseline Community Health Workers's attitude about physical activity promotion at 1 month | 1 month
Change from baseline Community Health Workers's attitude about physical activity promotion at 5 months | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Alex A Florindo, Ph.D., Principal Investigator — University of Sao Paulo
Locations (1):
- School of Arts, Sciences and Humanities, University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Florindo AA, Costa EF, Sa TH, dos Santos TI, Velardi M, Andrade DR. Physical activity promotion in primary health care in Brazil: a counseling model applied to community health workers. J Phys Act Health. 2014 Nov;11(8):1531-9. doi: 10.1123/jpah.2012-0260. Epub 2013 Dec 31. PMID 24385474
- See also: Research group website. — http://www.each.usp.br/gepaf/